CLINICAL TRIAL: NCT00740623
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Carisbamate as Adjunctive Therapy in Subjects With Partial Onset Seizures.
Brief Title: A Study of the Effectiveness, Safety, and Tolerability of Carisbamate as Add-On Therapy in Patients With Partial Onset Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015463; CARISEPY3013
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Epilepsy, Partial, Motor; Epilepsy, Complex Partial; Epilepsy, Simple Partial; Focal Motor Epilepsy
Keywords: Partial Onset Seizures; Simple Partial Seizures; Complex Partial Seizures
MeSH Terms: conditions — Epilepsy, Partial, Motor; Epilepsy, Complex Partial; Epilepsies, Partial; Seizures | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): Carisbamate 800 mg/day for 14 weeks
  Interventions: Drug: Carisbamate
- 002 (Experimental): Carisbamate 1,200 mg/day for 14 weeks
  Interventions: Drug: Carisbamate
- 003 (Placebo Comparator): placebo for 14 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Carisbamate — 800 mg/day for 14 weeks
  Arms: 001
Drug: placebo — placebo for 14 weeks
  Arms: 003
Drug: Carisbamate — 1,200 mg/day for 14 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety, and tolerability of carisbamate as add-on therapy for the treatment of partial onset seizures in patients with epilepsy.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), epilepsy afflicts more than 50 million people worldwide. Older antiepileptic drugs are still commonly used, despite a diverse range of side effects. New AEDs approved since the early 1990s have shown an improved tolerability profile. Nonetheless, approximately 30% of patients, particularly those with partial onset seizures, are not well controlled even on the newer treatments or they experience significant side effects secondary to treatment. Therefore, the development of new drugs with effectiveness or safety and tolerability advantages over currently marketed antiepileptic drugs is needed. This is a randomized (study medication assigned by chance), double-blind (neither the physician nor the patient knows the name of the assigned study medication), placebo-controlled, parallel-group, multicenter study. The study has 3 phases: an 8-week pretreatment phase including screening and a baseline period, a 14-week double blind treatment phase, including a 2-week titration period and a 12-week maintenance period, and a 4 week posttreatment phase. During the 56-day baseline period, patients will be required to have at least 6 partial onset seizures, no more than >= 100 partial onset seizures per 28 days, and no seizure-free period for more than 3 weeks to be eligible to enter the double-blind treatment phase of the study. During the double-blind treatment phase of study CARISEPY3013, patients will be randomly assigned to receive 800 mg/day carisbamate, 1,200 mg/day carisbamate, or placebo for 14 weeks. The total duration of study CARISEPY3013 is approximately 26 weeks for each subject. Patients who complete the double-blind treatment phase will be eligible to enter the separate extension study CARISEPY3014. Safety assessments include the monitoring of the frequency, severity, and timing of adverse events, clinical laboratory test results, 12-lead electrocardiogram (ECG) recordings, vital signs measurements, physical and neurologic examinations, the Physician Withdrawal Checklist for symptoms of withdrawal for those patients who taper and/or discontinue study drug, and pregnancy tests for females of childbearing potential. Assessments of effectiveness include seizure counts at every visit and the Quality of Life in Epilepsy-31 Patient Inventory questionnaire. A Medical Resource utilization questionnaire will be used to obtain cost-effectiveness information on carisbamate. The study hypothesis is that carisbamate is superior to placebo as add-on therapy (i.e., in addition to the current antiepileptic drugs that patients are taking) for the treatment of partial onset seizures in patients with epilepsy. Carisbamate 800 mg/day, 1,200 mg/day, or placebo taken twice daily in 2 equally divided doses, with or without food, and taken with noncarbonated water. A double-dummy design will be used so that all patients will take the same number of active drug and placebo tablets each day during the 14 weeks of the double blind treatment phase. Patients will continue to take a stable dosage or dosages of up to 3 antiepileptic drugs that they are already taking for their seizures during the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of partial onset seizures
* had a neuroimaging procedure (computed tomography [CT] or magnetic resonance imaging [MRI] within the past 5 years that excluded a progressive neurologic disorder
* History of inadequate response to at least 1 antiepileptic drug
* Current treatment with at least 1 and up to 3 antiepileptic drugs. To be eligible for the double-blind treatment phase of study CARISEPY3013, patients must: have at least 6 partial onset seizures during the 56-day baseline period
* Have not had > = 100 partial onset seizures per 28 days in the baseline period
* And no seizure-free period of more than 3 weeks during the baseline period.

Exclusion Criteria:

* History of status epilepticus or epilepsia partialis continua in the 6 months before study entry
* Have a generalized epileptic syndrome
* have a diagnosis of Lennox-Gastaut Syndrome
* Currently experiencing seizures that cannot be counted accurately
* have experienced rates of > = 100 partial onset seizures in any monthly period in the 6 months before study entry
* Have a history of any current or past nonepileptic seizures, including psychogenic seizures
* History of or current serious or medically unstable systemic disease
* evidence of cardiac disease, including unstable angina, myocardial infarction, within the past 2 years, uncontrolled heart failure, major arrhythmias, congenital short QT syndrome, or significant shortening or lengthening of the QTc interval of the electrocardiogram
* progressive neurologic disorder, such as a brain tumor, demyelinating disease, and degenerative CNS disease, or active CNS infection
* current or past (within the past year) major psychotic disorder
* History of suicidal or homicidal ideation within the past 2 years, or an episode of suicide attempt or homicide at any time in the past.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoints are percent reduction in partial onset seizure frequency in the US and the rest of the world (excluding Europe, Australia, New Zealand, S Africa), and responder rate for Europe, Australia, New Zealand, S Africa | from baseline relative to the entire double-blind treatment phase (14 weeks)

SECONDARY OUTCOMES:
Secondary endpoints are percent reduction in partial onset seizure frequency for EuropeAustraliaNew Zealand S Africa, percent reduction in secondarily generalized seizure and time to onset of treatment effect on partial onset seizure frequency reduction | from baseline relative to the entire double-blind treatment phase (14 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Lu C, Zheng J, Cao Y, Bresnahan R, Martin-McGill KJ. Carisbamate add-on therapy for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD012121. doi: 10.1002/14651858.CD012121.pub2. PMID 34870321
- [Derived] Halford JJ, Ben-Menachem E, Kwan P, Ness S, Schmitt J, Eerdekens M, Novak G. A randomized, double-blind, placebo-controlled study of the efficacy, safety, and tolerability of adjunctive carisbamate treatment in patients with partial-onset seizures. Epilepsia. 2011 Apr;52(4):816-25. doi: 10.1111/j.1528-1167.2010.02960.x. Epub 2011 Feb 14. PMID 21320109